CLINICAL TRIAL: NCT02385578
Title: An Educational Intervention, the First Step of the Train the Trainer (TTT) Plan, to Improve the Young Endoscopist's Ability to Find the Early Gastric Cancer:Prospective Study With Historical Control
Brief Title: the Train the Trainer (TTT) Plan, to Improve the Young Endoscopist's Ability to Find the Early Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: B2015-048
Record Dates: First submitted 2015-02-28; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Early Gastric Cancer
Keywords: VS (vessel plus surface) classification system; Magnified endoscopy with narrow band imaging (ME-NBI); the rate of detection
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The control group (No Intervention): no intervention
- The experimental group (Experimental): an educational intervention
  Interventions: Other: an educational intervention

INTERVENTIONS:
Other: an educational intervention — the first step of the train the trainer plan(TTT) ,which including the diagnosis and operation "hand in hand" teach by Professor Yano Takeshiin,and the case discussion,and so on
  Other Names: the first step of the train the trainer plan(TTT)
  Arms: The experimental group

SUMMARY:
AIM Verified if the first stage of the Train the trainer (TTT)plan could improve the young endoscopist's ability to detect the early gastric cancer（EGC）.

METHOD

1. a retrospective analysis of the ten young endoscopist's painless gastroscopy examination from January 1, 2014 to December 31, 2014. According mainly to the endoscopic report and pateint's History, quantity of gastroscope, gastric cancer and the early gastric cancer.
2. the first step of the train the trainer plan(TTT) activised in March 19-20,2015,which including the diagnosis and operation "hand in hand" teach by Professor Yano Takeshiin,and the case discussion,and so on. Five young endoscopist accepted the TTT plan and the other five not accepted.
3. The five doctors who accepted the TTT do the gastroendoscopy in accordance with the TTT content (for the T1 period),.(1) the patient's name, (2)gender, (3)age,(4)past medical history (Helicobacter pylori<HP>, gastritis, gastric ulcer, oral drug operation, etc.),（5）gastroscope operation time,(6)the location of the lesion- longitudinal (upper, middle and lower),(7) the location of the lesion -circumferential (lessor curvature, Greater curvature, anterior wall, posterior wall),(8) lesion size, (9)conventional white-light imaging (red, white, no change), (10)magnifying endoscopy with narrow-band imaging (EM-NBI) microvascular and mirosurface pattern VS classification system(VSCS) (boundaries, microvascular pattern and microsurface pattern; don't do it), (11)microscopy types (uplift type, flat type, concave type or IIc I/IIa or IIb), (12)histological type (differentiated and undifferentiated type) and (13) pathological (low grade neoplasia, high-level neoplasia etc.). For the treatment of endoscopy submucosal dissection (ESD) patients, further pathological results were recorded after ESD, including the pathology, edge and basal conditions. The other five doctors do the gastroendoscopy as they do before. (300 cases / person)
4. 2-4 TTT activity ;The five doctors who accepted the TTT do the gastroendoscopy in accordance with the TTT content (for the T2-T4 period),.The other five doctors do the gastroendoscopy as they do before.
5. Statistics the number of early gastric cancer have been found by the five young doctors, and how mang gastroscopy they have done.pay attention to The rates of EGC detection.

DETAILED DESCRIPTION:
AIM Verified if the first stage of the Train the trainer (TTT)plan could improve the young endoscopist's ability to detect the early gastric cancer.

GROUP The control group five young endoscopist not accepted the TTT The experimental group five young endoscopist accepted the TTT CRITERIA The entry criteria (A) retrospective part (1) The gastroscopy patients was operated by the ten doctors in 2014: (2) painless gastroscopy(intravenous anesthesia); (3) age: 18-70 years old; male or female (B): prospective part

(1) consistent with gastroscopy indications: (2) painless gastroscopy(intravenous anesthesia); (3) age: 18-70 years old; male or female (4) signed the informed consent.

Exclusion criteria ( retrospective part and prospective part)

1. those patients who underwent gastrectomy
2. the emergency gastroscopy, such as, esophageal foreign body, gastric foreign body, upper gastrointestinal hemorrhage. ;
3. serious gastric hemorrhage or food residue that influence endoscopist's observation;
4. those had been diagnosed outside the hospital before gastroscopy this time;
5. those took oral anticoagulants and can't do biopsy examination;
6. those were not suitable for endoscopic contraindication for endoscopic examination or endoscopic biopsy;
7. do not fit into the experiment;
8. don't do as the test plan demand.

METHOD

1. a retrospective analysis of the ten young endoscopist's painless gastroscopy examination from January 1, 2014 to December 31, 2014. According mainly to the endoscopic report and pateint's History, quantity of gastroscope, gastric cancer and the early gastric cancer. In addition, for early gastric cancer patients, it was record,(1) the patient's name, (2)gender, (3)age, (4)the location of the lesion- longitudinal (upper, middle and lower),(5) the location of the lesion -circumferential (lessor curvature, Greater curvature, anterior wall, posterior wall),(6) lesion size, (7)conventional white-light imaging (red, white, no change), (8)EM-NBI VS type (boundaries, microvascular pattern and microsurface pattern; don't do it), (9)microscopy types (uplift type, flat type, concave type or IIc I/IIa or IIb), (10)histological type (differentiated and undifferentiated type) and (11) pathological (low grade neoplasia, high-level neoplasia etc.). For the treatment of ESD patients, further pathological results were recorded after ESD, including the pathology, edge and basal conditions.

   Note:

   (A) those had been diagnosed outside the hospital before gastroscopy, withhold, listed separately.

   (B) for anesthesia, or not to determine whether anesthesia, withhold, separately listed; (C) considering the actual clinical situation, in the absence of pathological report, endoscopy reports generally will not report "early gastric cancer", but will use descriptive language diagnosis as "erosion" "apophysis" " ulcer". The investigators will find out the suspected early gastric cancer, then go on to confirm the diagnosis by the pathologic findings.

   (D) considering the actual clinical situation, the investigators often wrote the Malignant tumor （MT） instead of the gastric cancer in patients' report. Don't miss the descriptive language as "ulcer" patients. Found out the suspected patients and confirmed by pathology.
2. the first step of the train the trainer plan(TTT) activised in March 19-20,2015,which including the diagnosis and operation "hand in hand" teach by Professor Yano Takeshiin,and the case discussion,and so on. Core: First, a detailed examination by white light is used to look for an irregular margin or a depressed spiny area.Then narrow-band imaging is used to look for a demarcation line, an microvascular pattern and microsurface pattern .five young endoscopist accepted the TTT plan and the other five not accepted.
3. The five doctors who accepted the TTT do the gastroendoscopy in accordance with the TTT content (for the T1 period),.(1) the patient's name, (2)gender, (3)age,(4)past medical history (HP, gastritis, gastric ulcer, oral drug operation, etc.),（5）gastroscope operation time,(6)the location of the lesion- longitudinal (upper, middle and lower),(7) the location of the lesion -circumferential (lessor curvature, Greater curvature, anterior wall, posterior wall),(8) lesion size, (9)conventional white-light imaging (red, white, no change), (10)EM-NBI VS type (boundaries, microvascular pattern and microsurface pattern; don't do it), (11)microscopy types (uplift type, flat type, concave type or IIc I/IIa or IIb), (12)histological type (differentiated and undifferentiated type) and (13) pathological (low grade neoplasia, high-level neoplasia etc.). For the treatment of ESD patients, further pathological results were recorded after ESD, including the pathology, edge and basal conditions. The other five doctors do the gastroendoscopy as they do before. (300 cases / person)
4. second TTT activity (2015 July -8 months),;
5. The five doctors who accepted the TTT do the gastroendoscopy in accordance with the TTT content (for the T2 period),.The other five doctors do the gastroendoscopy as they do before. (300 cases / person)
6. third TTT activity (2015 November -12 months);
7. The five doctors who accepted the TTT do the gastroendoscopy in accordance with the TTT content (for the T3 period),The other five doctors do the gastroendoscopy as they do before. (300 cases / person)
8. fourth TTT activity (2016 February -3 months);
9. The five doctors who accepted the TTT do the gastroendoscopy in accordance with the TTT content (for the T4 period),The other five doctors do the gastroendoscopy as they do before. (300 cases / person)
10. Statistics the number of early gastric cancer have been found by the five young doctors, and how mang gastroscopy they have done.

(A) List the general condition of patients before and after TTT; found the location of the tumor, whether the same type? (B) The rates of EGC detection before and after the TTT? Is the rates of Gastric cancer(GC) detection increasing? (C)The rates of EGC detection between the doctor accepted the TTT and not? (D) is the rates of EGC detection different among T1, T2, T3, T4 ? Is the rates of Gastric cancer detection increasing? (F) early cancer patients was found after TTT training, comparison the endoscopic diagnosis with Pathology, and pay attention to accuracy, sensitivity, false positive rate and false negative rate （ME-NBI）. And the reason analysis.

ELIGIBILITY:
Inclusion Criteria:

(A) retrospective part (1) The gastroscopy patients was operated by the ten doctors in 2014: (2) painless gastroscopy(intravenous anesthesia) (3) age: 18-70 years old; male or female ( - prospective part

1. consistent with gastroscopy indications:
2. painless gastroscopy(intravenous anesthesia)
3. age: 18-70 years old; male or female
4. signed the informed consent.

Exclusion Criteria:

( retrospective part and prospective part)

1. those patients who underwent gastrectomy
2. the emergency gastroscopy, such as, esophageal foreign body, gastric foreign body, upper gastrointestinal hemorrhage. ;
3. serious gastric hemorrhage or food residue that influence endoscopist's observation;
4. those had been diagnosed outside the hospital before gastroscopy this time;
5. those took oral anticoagulants and can't do biopsy examination;
6. those were not suitable for endoscopic contraindication for endoscopic examination or endoscopic biopsy;
7. do not fit into the experiment;
8. don't do as the test plan demand. -

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16000 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The rates of EGC detection | 16 months
  The rates of EGC detection before and after the TTT in the experiment group or in the control group? The rates of EGC detection between the experiment group and the control group after TTT

CONTACTS AND LOCATIONS:
Overall Officials: Yao li-qing, MD, Principal Investigator — Shanghai Zhongshan Hospital

REFERENCES:
- [Result] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Result] Suvakovic Z, Bramble MG, Jones R, Wilson C, Idle N, Ryott J. Improving the detection rate of early gastric cancer requires more than open access gastroscopy: a five year study. Gut. 1997 Sep;41(3):308-13. doi: 10.1136/gut.41.3.308. PMID 9378383
- [Result] Kanesaka T, Sekikawa A, Tsumura T, Maruo T, Osaki Y, Wakasa T, Shintaku M, Yao K. Absent microsurface pattern is characteristic of early gastric cancer of undifferentiated type: magnifying endoscopy with narrow-band imaging. Gastrointest Endosc. 2014 Dec;80(6):1194-1198.e1. doi: 10.1016/j.gie.2014.08.021. Epub 2014 Oct 16. No abstract available. PMID 25442093
- [Result] Mabe K, Yao K, Nojima M, Tanuma T, Kato M. An educational intervention to improve the endoscopist's ability to correctly diagnose small gastric lesions using magnifying endoscopy with narrow-band imaging. Ann Gastroenterol. 2014;27(2):149-155. PMID 24733047
- [Result] Yao K, Doyama H, Gotoda T, Ishikawa H, Nagahama T, Yokoi C, Oda I, Machida H, Uchita K, Tabuchi M. Diagnostic performance and limitations of magnifying narrow-band imaging in screening endoscopy of early gastric cancer: a prospective multicenter feasibility study. Gastric Cancer. 2014 Oct;17(4):669-79. doi: 10.1007/s10120-013-0332-0. Epub 2014 Jan 10. PMID 24407989
- [Result] Kanemitsu T, Yao K, Nagahama T, Fujiwara S, Takaki Y, Ono Y, Matsushima Y, Matsui T, Tanabe H, Ota A, Iwashita A. The vessels within epithelial circle (VEC) pattern as visualized by magnifying endoscopy with narrow-band imaging (ME-NBI) is a useful marker for the diagnosis of papillary adenocarcinoma: a case-controlled study. Gastric Cancer. 2014;17(3):469-77. doi: 10.1007/s10120-013-0295-1. Epub 2013 Sep 15. PMID 24037102
- [Result] Yao K. The endoscopic diagnosis of early gastric cancer. Ann Gastroenterol. 2013;26(1):11-22. PMID 24714327
- [Result] Zhang Q, Chen ZY, Chen CD, Liu T, Tang XW, Ren YT, Huang SL, Cui XB, An SL, Xiao B, Bai Y, Liu SD, Jiang B, Zhi FC, Gong W. Training in early gastric cancer diagnosis improves the detection rate of early gastric cancer: an observational study in China. Medicine (Baltimore). 2015 Jan;94(2):e384. doi: 10.1097/MD.0000000000000384. PMID 25590840